CLINICAL TRIAL: NCT00720382
Title: Active Controlled Trial of the Safety and Tolerability of MP 03-036 (Astepro 0.15%) in Patients With Perennial Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Tolerability of a Nasal Spray to Treat Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP436
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — azelastine; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 0.15% azelastine hydrochloride 1644 mcg
  Interventions: Drug: 0.15% azelastine hydrochloride
- 2 (Experimental): Mometasone furoate 200 mcg
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: 0.15% azelastine hydrochloride — 1644 mcg (205.5 mcg/spray) 2 sprays per nostril twice a day/AM and PM
  Arms: 1
Drug: Mometasone furoate — 200 mcg (50 mcg/spray) 2 sprays per nostril Once a day (AM)
  Arms: 2

SUMMARY:
The purpose of this study is to determine if one allergy treatment (0.15% azelastine hydrochloride) is as safe as mometasone furoate (nasonex) alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 years and older with a compatible history greater than or equal to 1 year of rhinitis due to perennial allergies.
* Must be willing and able to provide informed consent and to participate in all study procedures
* Must be in generally good health
* Positive skin test to a prevalent perennial allergen

Exclusion Criteria:

* On nasal examination, the presence of nasal mucosal erosion, nasal ulceration or nasal septal perforation
* Use of any investigational drug within 30 days of the first visit
* Any nasal surgery or sinus surgery within the previous year
* Presence of any hypersensitivity to drugs similar to azelastine or mometasone furoate and to either sorbital or sucralose
* Women who are pregnant or nursing
* Women who are not using an acceptable method of birth control
* Nasal Diseases likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa or clinically significant nasal polyposis or nasal structural abnormalities.
* Asthma or other lung diseases such as COPD. Mild asthma symptoms may be considered after consultation with investigator.
* Patients with Arrythmia
* Patients with know history of alcohol and drug abuse
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor, might significantly alter the evaluation of the study.
* Use of medications that could affect the study results

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M. Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (59):
- United States (59):
  - Center of Research Excellence, LLC, Oxford, Alabama
  - AABI Associates Medical Group, Fountain Valley, California
  - Allergy and Asthma Specialist Medical Group, Huntington Beach, California
  - West Coast Clinical Trials, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Cntr, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - Allergy and Asthma Care of Florida, Ocala, Florida
  - Allergy and Asthma DTC, Tallahassee, Florida
  - Georgia Pollens Clinical Research Centers Inc, Albany, Georgia
  - Aeroallergy Research Laboratories of Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - RX R+D, Metairie, Louisiana
  - Institute for Asthma and Allergy PC, Wheaton, Maryland
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Allergy and Asthma Research NJ inc, Mount Laurel, New Jersey
  - Atlantic Research Center, Ocean City, New Jersey
  - Dr. Perin, Teaneck, New Jersey
  - Medical Research Associates of CNY, PLLC, North Syracuse, New York
  - AAIR Research Center, Rochester, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - New Horizon's Clinical Research, Cincinnati, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical, Edmond, Oklahoma
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy Asthma and Dermatology Research, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy and Asthma Specialist PC, Blue Bell, Pennsylvania
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - Asthma, Nasal Disease & Allergy Research Center of New England, Providence, Rhode Island
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - Allergy and Asthma Associates, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - SWAAA Research Center, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Live Oak Allergy and Asthma Clinic, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - VA Adult and Pediatric Allergy and Asthma, Richmond, Virginia
  - Asthma, Inc., Seattle, Washington
  - Advanced Healthcare, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Bousquet J, Klimek L, Kuhl HC, Nguyen DT, Kumar Ramalingam R, Canonica GW, Berger WE. In perennial allergic rhinitis, RQLQ is improved similarly by Azelastine 0.15 and mometasone furoate. World Allergy Organ J. 2025 Jan 8;18(1):101021. doi: 10.1016/j.waojou.2024.101021. eCollection 2025 Jan. PMID 39885937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First observation: 09 MAR 2007 Last observation: 20 JUN 2008
Pre-assignment Details: Subjects participated in a 7 day screening period to identify appropriate subjects based on symptom scores.
Groups:
- Astepro 0.15%: 0.15% azelastine hydrochloride 1644 mcg
- Nasonex®: Mometasone furoate 200 mcg
Period: Overall Study
Arm/Group | Astepro 0.15% | Nasonex®
Started | 466 | 237
Completed | 290 | 178
Not Completed | 176 | 59
Not completed — Adverse Event | 54 | 17
Not completed — Lack of Efficacy | 18 | 7
Not completed — Non-Compliance | 15 | 5
Not completed — Withdrawal by Subject | 47 | 11
Not completed — Lost to Follow-up | 28 | 14
Not completed — administrative | 14 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Astepro 0.15% | Nasonex® | Total
Number analyzed (Participants) | 466 | 237 | 703
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 18 | 55
  Between 18 and 65 years | 410 | 211 | 621
  >=65 years | 19 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (14.54) | 39.1 (14.61) | 39.2 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310 | 175 | 485
  Male | 156 | 62 | 218
Region of Enrollment [Number; unit: participants]
  United States | 466 | 237 | 703

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Direct Visual Nasal Exams to 12 Months
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa. Nasal irritation was rated: 0 = None, Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion, Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: Change from baseline to 12 months
Measure: Number; unit: Participants
Arm/Group | Astepro 0.15% | Nasonex®
Number analyzed (Participants) | 466 | 237
Participants
  Epistaxis - Day 1 | 466 | 237
  None | 456 | 229
  Mild | 10 | 8
  Moderate | 0 | 0
  Severe | 0 | 0
  Epistaxis - Month 12/ET | 402 | 220
  None | 387 | 213
  Mild | 15 | 7
  Moderate | 0 | 0
  Severe | 0 | 0
  Nasal Irritation - Day 1 | 466 | 237
  None | 425 | 217
  Grade 1A | 37 | 17
  Grade 1B | 2 | 3
  Grade 2 | 2 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Nasal Irritation - Month 12/ET | 402 | 220
  None | 374 | 200
  Grade 1A | 22 | 17
  Grade 1B | 4 | 2
  Grade 2 | 2 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 1
  Conjunctival injection - Day 1 | 466 | 237
  None | 340 | 164
  Mild | 100 | 58
  Moderate | 24 | 14
  Severe | 2 | 1
  Conjunctival injection - Month 12/ET | 402 | 220
  None | 336 | 182
  Mild | 56 | 31
  Moderate | 8 | 7
  Severe | 2 | 0
  Erythematous TM - Day 1 | 466 | 236
  None | 443 | 226
  Mild | 21 | 8
  Moderate | 2 | 1
  Severe | 0 | 1
  Erythematous TM - Month 12/ET | 402 | 220
  None | 392 | 206
  Mild | 9 | 12
  Moderate | 1 | 2
  Severe | 0 | 0
  Lymphadenophthy-Day 1 | 465 | 237
  None | 433 | 225
  Mild | 30 | 12
  Moderate | 2 | 0
  Severe | 0 | 0
  Lymphadenopathy - Month 12/ET | 402 | 220
  None | 388 | 210
  Mild | 13 | 9
  Moderate | 1 | 1
  Severe | 0 | 0
  Mucosal Edema - Day 1 | 466 | 237
  None | 92 | 42
  Mild | 162 | 87
  Moderate | 181 | 96
  Severe | 31 | 12
  Mucosal Edema - Month 12/ET | 402 | 220
  None | 101 | 54
  Mild | 157 | 94
  Moderate | 129 | 66
  Severe | 15 | 6
  Nasal Discharge - Day 1 | 466 | 237
  None | 178 | 89
  Mild | 202 | 110
  Moderate | 78 | 33
  Severe | 8 | 5
  Nasal Discharge - Month 12/ET | 402 | 220
  None | 182 | 90
  Mild | 163 | 107
  Moderate | 53 | 22
  Severe | 4 | 1
  Mucosal Erythema - Day 1 | 466 | 237
  None | 258 | 145
  Mild | 153 | 67
  Moderate | 54 | 21
  Severe | 1 | 4
  Mucosal Erythema - Month 12/ET | 402 | 220
  None | 254 | 142
  Mild | 114 | 58
  Moderate | 31 | 20
  Severe | 3 | 0
  Mucosal Bleeding - Day 1 | 466 | 237
  None | 451 | 224
  Mild | 15 | 11
  Moderate | 0 | 1
  Severe | 0 | 1
  Mucosal Bleeding - Month 12/ET | 402 | 220
  None | 384 | 208
  Mild | 17 | 11
  Moderate | 1 | 1
  Severe | 0 | 0
  Crusting of Mucosa - Day 1 | 466 | 237
  None | 412 | 215
  Mild | 46 | 20
  Moderate | 8 | 1
  Severe | 0 | 1
  Crusting of Mucosa - Month 12/ET | 402 | 220
  None | 373 | 197
  Mild | 20 | 22
  Moderate | 9 | 1
  Severe | 0 | 0

2. Other Pre Specified Outcome: Change From Baseline to 12 Months in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Compared to Placebo in Subjects 18 Years of Age and Older
Description: A 28-item RQLQ was completed on Day 1, Month 1, Month 3, Month 6, month 9 and month 12 or Early termination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time.
  Domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: change from baseline to 12 months
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Astepro 0.15% | Nasonex®
Number analyzed (Participants) | 466 | 237
Units on a scale
  Overall Score Baseline | 2.78 (1.227) | 2.75 (1.191)
  Month 1 | -0.97 (1.201) | -0.97 (1.245)
  Month 3 | -1.15 (1.256) | -1.27 (1.379)
  Month 6 | -1.13 (1.236) | -1.29 (1.372)
  Month 9 | -1.17 (1.219) | -1.31 (1.425)
  Month 12/ET | -0.90 (1.302) | -1.11 (1.364)
Statistical Analysis 1: Comparison: Astepro 0.15% vs Nasonex®; Overall baseline score; Test type: Superiority or Other; p = 0.783, ANCOVA; ANCOVA was used as a model containing treatment group and site as fixed effects with the baseline value used as covariate
Statistical Analysis 2: Comparison: Astepro 0.15% vs Nasonex®; Change from baseline to Month 1; Test type: Superiority or Other; p = 0.971, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Astepro 0.15% vs Nasonex®; Change from baseline to Month 3; Test type: Superiority or Other; p = 0.206, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Astepro 0.15% vs Nasonex®; Change from baseline to Month 6; Test type: Superiority or Other; p = 0.111, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Astepro 0.15% vs Nasonex®; Change from baseline to Month 9; Test type: Superiority or Other; p = 0.181, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Astepro 0.15% vs Nasonex®; Change from Baseline to Month 12/Early Term; Test type: Superiority or Other; p = 0.037, ANCOVA; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Ae's greater than 2% in MP03-36 (Astepro 0.15%). Any significant findings found on the nasal exams were reported as AE's and would be found here.
Arm/Group | Astepro 0.15% | Nasonex®
Serious Adverse Events (participants affected / at risk) | 4/466 | 4/237
Other Adverse Events (participants affected / at risk) | 349/466 | 163/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astepro 0.15% (N=466) | Nasonex® (N=237)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astepro 0.15% (N=466) | Nasonex® (N=237)
DYSGEUSIA (Nervous system disorders) | 62 (62) | 3 (3)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 46 (46) | 19 (19)
SINUSITIS (Infections and infestations) | 44 (44) | 19 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 43 (43) | 28 (28)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 43 (43) | 24 (24)
NASOPHARYNGITIS (Infections and infestations) | 43 (43) | 20 (20)
HEADACHE (Nervous system disorders) | 41 (41) | 30 (30)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 14 (14)
BRONCHITIS (Infections and infestations) | 19 (19) | 6 (6)
FATIGUE (General disorders) | 19 (19) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 17 (17) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 (16) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 12 (12)
INFLUENZA (Infections and infestations) | 15 (15) | 9 (9)
SINUS HEADACHE (Nervous system disorders) | 15 (15) | 4 (4)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 0 (0)
MUCOSAL EROSION (General disorders) | 13 (13) | 6 (6)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. Authorship will be determined by mutual agreement.